CLINICAL TRIAL: NCT00652353
Title: Efficacy of a Mnemonic to Improve Knowledge of the Ottawa Ankle and Foot Rules Among Medical Students and Residents; a Randomized Controlled Trial.
Brief Title: Mnemonic for the Ottawa Ankle Rule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 44-55-66-PM
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Ankle Trauma; Education
Keywords: Clinical decision rule; Ottawa Ankle Rule; Ottawa Foot Rule; Ankle; Trauma; Education; Foot Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will be given a standardized information sheet providing a mnemonics to help remember the Ottawa Ankle and foot Rules.
  Interventions: Other: 44-55-66-PM
- 0 (Placebo Comparator): control group
  Interventions: Other: control

INTERVENTIONS:
Other: 44-55-66-PM — The mnemonic 44-55-66-PM helps to remember the components of the Ottawa Ankle and foot Rule.
  44: Is to remember that an X-ray is required if the patients is unable to walk 4 steps at the moment of the Accident AND during the physical examination 55: Is to remember that an X-ray of the foot is required if the patient has pain at the basis of the 5Th metatarsal of at the 5caphoid 66-PM: Is to remember that an X-ray of the ankle is required if the patient has pain in the Posterior of the lateral or medial malleolar
  Arms: Intervention
Other: control — Participants will be instructed of the components of the Ottawa Ankle Rule on a standardized sheet
  Arms: 0

SUMMARY:
The purpose of this study is to evaluate wether the use of a mnemonic strategy could improve the recall of the Ottawa Ankle and foot Rules' guidelines among medical students and residents

ELIGIBILITY:
Inclusion Criteria:

* Being a medical student in rotation in pediatrics at CHU Sainte-Justine
* Being a resident in pediatric emergency rotation at CHU Sainte-Justine

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Knowledge of the components of the Ottawa Ankle rule based on a 13 points evaluation | 3-4 weeks after intervention
Knowledge of the components of the Ottawa foot rule based on a 10 points evaluation | 3-4 weeks

SECONDARY OUTCOMES:
Proportion of perfect knowledge of the Ottawa Ankle and Foot Rules | 3-4 weeks
Score on an exam evaluating management of 20 case scenarios describing patients with an ankle or foot trauma | 3-4 weeks post intervention
Knowledge of the 13 components of the Ottawa Ankle Rule and the 10 components of the Ottawa Foot Rule | 6 months post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Result] Gravel J, Roy M, Carriere B. 44-55-66-PM, a mnemonic that improves retention of the Ottawa Ankle and Foot Rules: a randomized controlled trial. Acad Emerg Med. 2010 Aug;17(8):859-64. doi: 10.1111/j.1553-2712.2010.00731.x. PMID 20670323